CLINICAL TRIAL: NCT03159910
Title: Reducing Shoulder Complaints in Employees With High Occupational Shoulder Exposures: a Cluster-randomised Controlled Study (The Shoulder-Café Study)
Brief Title: Reducing Shoulder Complaints in Employees With High Occupational Shoulder Exposures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: Regional Hospital West Jutland (Other); Aarhus University Hospital (Other); University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JutlandRH
Record Dates: First submitted 2017-05-11; First posted 2017-05-19 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2019-09

CONDITIONS: Shoulder Pain
Keywords: Shoulder Pain; Occupational Exposure; Clinical Trial
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be masked with respect to mechanical shoulder exposures. Statistical analyses will be performed blinded to intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder-Café (intervention) (Experimental): A Shoulder-Café intervention consists of three café-meetings.
  Interventions: Behavioral: Shoulder-Café
- Shoulder-Guidance (control) (Active Comparator): The Shoulder-Guidance intervention consists of an initial individual appointment and two e-mail contacts.
  Interventions: Behavioral: Shoulder-Guidance

INTERVENTIONS:
Behavioral: Shoulder-Café — Education and individual counselling, clinical examination, supervised shoulder exercise. Some participants can be offered a workplace visit.
  Arms: Shoulder-Café (intervention)
Behavioral: Shoulder-Guidance — Home-based shoulder exercise and written counselling.
  Arms: Shoulder-Guidance (control)

SUMMARY:
Aim: To evaluate the effectiveness of Shoulder-Café (intervention) compared to Shoulder-Guidance (control intervention) with respect to shoulder exposures and shoulder complaints.

Hypothesis: The Shoulder-Café, which unifies education, diagnostic clarification, supervised and home-based shoulder exercises, and advice from a health and safety consultant on workplace interventions, will reduce shoulder exposures and shoulder complaints more effectively than an individual-oriented control intervention with home-based shoulder exercises and written general advice on workplace interventions.

DETAILED DESCRIPTION:
Introduction:

Shoulder complaints prevail in the working age population and constitute a common cause of contacts with general practitioners. In occupations with high mechanical shoulder exposures, these complaints are especially frequent. Persons with high occupational mechanical shoulder exposures and shoulder complaints seem an obvious target group for secondary prevention efforts, and more research on interventions targeting shoulder complaints in occupations with high shoulder exposures is needed.

The aim is to develop and evaluate a Shoulder-Café intervention to reduce high occupational mechanical shoulder exposures and prolonged shoulder complaints.

The specific objectives are:

I. To evaluate the effectiveness of the Shoulder-Café as compared to the control-intervention, the Shoulder-Guidance, measured on reductions in shoulder complaints.

II. To evaluate the effectiveness of the Shoulder-Café as compared to the Shoulder-Guidance measured on reductions in occupational mechanical shoulder exposures.

III. To identify the influence of shoulder exercises and reduced occupational mechanical shoulder exposures, respectively, on shoulder complaints.

The hypothesis is that the Shoulder-Café will reduce shoulder exposures and shoulder complaints more effectively than the Shoulder-Guidance. Furthermore, a hypothesis is that fear avoidance beliefs is reduced and the degree to which the participants feel informed about the nature of their complaints and their remedies is increased more effectively with the Shoulder-Café compared to the control intervention.

Method:

The project consists of a two-armed, cluster-randomised controlled trial with randomisation at company level (objectives I and II) and a prospective cohort study based on the cluster-randomised study (objective III).

Follow-up: A questionnaire 3 and 9 months after end of intervention with e.g. OSS.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Employed in occupations with expected high mechanical shoulder exposures (industry, construction and service)
* Shoulder complaints
* Able to read and understand Danish

Exclusion Criteria:

* Previous shoulder surgery
* Breast cancer operation
* Pregnancy
* Sickness absence expected to continue into the intervention period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Shoulder complaints | Follow-up 3 months after end of intervention.
  Monitored with the Danish version of the Oxford Shoulder Score (questionnaire).
Mechanical shoulder exposures | Follow-up at end of intervention, an average of 2-3 months
  Measured during 1-5 working days in terms of % time with the arm elevated at different angles and shoulder angular velocity (°/s) using an Axivity accelerometer. Degree of exertion for the arms monitored with Borg CR10 (questionnaire). Participants will fill out questions in Borg CR 10 when they are using the Axivity accelerometer.

SECONDARY OUTCOMES:
Fear Avoidance Beliefs (FABQ) about physical activity (PA) | Follow-up 3 and 9 months after end of intervention.
  Monitored with FABQ-PA in a version modified to the shoulder (questionnaire)
Patients' Global Impression of Change | Follow-up 3 months after end of intervention.
  Measured on a 7 point Likert scale.
Shoulder complaints | Follow-up 9 months after end of intervention
  Monitored with the Danish version of the Oxford Shoulder Score

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Trøstrup, MsC, Principal Investigator — Elective Surgery Centre, Silkeborg Regional Hospital, Regional Hospital Central Jutland.
Locations (1):
- Elective Surgery Centre, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frich LH, Noergaard PM, Brorson S. Validation of the Danish version of Oxford Shoulder Score. Dan Med Bull. 2011 Nov;58(11):A4335. PMID 22047932
- [Background] Schmidt S, Ferrer M, Gonzalez M, Gonzalez N, Valderas JM, Alonso J, Escobar A, Vrotsou K; EMPRO Group. Evaluation of shoulder-specific patient-reported outcome measures: a systematic and standardized comparison of available evidence. J Shoulder Elbow Surg. 2014 Mar;23(3):434-44. doi: 10.1016/j.jse.2013.09.029. Epub 2014 Jan 7. PMID 24406123
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Mintken PE, Cleland JA, Whitman JM, George SZ. Psychometric properties of the Fear-Avoidance Beliefs Questionnaire and Tampa Scale of Kinesiophobia in patients with shoulder pain. Arch Phys Med Rehabil. 2010 Jul;91(7):1128-36. doi: 10.1016/j.apmr.2010.04.009. PMID 20599053
- [Background] Borg G. Psychophysical scaling with applications in physical work and the perception of exertion. Scand J Work Environ Health. 1990;16 Suppl 1:55-8. doi: 10.5271/sjweh.1815. PMID 2345867
- [Background] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Background] Virta L, Joranger P, Brox JI, Eriksson R. Costs of shoulder pain and resource use in primary health care: a cost-of-illness study in Sweden. BMC Musculoskelet Disord. 2012 Feb 10;13:17. doi: 10.1186/1471-2474-13-17. PMID 22325050
- [Background] Mitchell C, Adebajo A, Hay E, Carr A. Shoulder pain: diagnosis and management in primary care. BMJ. 2005 Nov 12;331(7525):1124-8. doi: 10.1136/bmj.331.7525.1124. No abstract available. PMID 16282408
- [Background] van Rijn RM, Huisstede BM, Koes BW, Burdorf A. Associations between work-related factors and specific disorders of the shoulder--a systematic review of the literature. Scand J Work Environ Health. 2010 May;36(3):189-201. doi: 10.5271/sjweh.2895. Epub 2010 Jan 22. PMID 20094690
- [Background] Anton D, Mizner RL, Hess JA. The effect of lift teams on kinematics and muscle activity of the upper extremity and trunk in bricklayers. J Orthop Sports Phys Ther. 2013 Apr;43(4):232-41. doi: 10.2519/jospt.2013.4249. Epub 2013 Jan 14. PMID 23321695
- [Background] Rempel D, Star D, Barr A, Blanco MM, Janowitz I. Field evaluation of a modified intervention for overhead drilling. J Occup Environ Hyg. 2010 Apr;7(4):194-202. doi: 10.1080/15459620903558491. PMID 20094939
- [Derived] Trostrup J, Frost P, Dalboge A, Mikkelsen LR, Hoybye MT, Jorgensen LB, Casper SD, Klebe TM, Svendsen SW. Reducing Shoulder Complaints in Employees with High Occupational Shoulder Exposures: A Cluster-Randomised Controlled Study (The Shoulder-Cafe Study). J Occup Rehabil. 2023 Sep;33(3):473-485. doi: 10.1007/s10926-022-10086-z. Epub 2022 Dec 13. PMID 36512271
- [Derived] Trostrup J, Svendsen SW, Dalboge A, Mikkelsen LR, Hoybye MT, Jorgensen LB, Klebe TM, Frost P. Increased shoulder pain across an exercise session and subsequent shoulder exercise: a prospective cohort study. BMC Musculoskelet Disord. 2022 Jul 29;23(1):726. doi: 10.1186/s12891-022-05674-2. PMID 35906579
- [Derived] Trostrup J, Mikkelsen LR, Frost P, Dalboge A, Hoybye MT, Casper SD, Jorgensen LB, Klebe TM, Svendsen SW. Reducing shoulder complaints in employees with high occupational shoulder exposures: study protocol for a cluster-randomised controlled study (The Shoulder-Cafe Study). Trials. 2019 Nov 12;20(1):627. doi: 10.1186/s13063-019-3703-y. PMID 31718683